CLINICAL TRIAL: NCT00956644
Title: Efficacy and Safety of Irbesartan/Amlodipine Fixed Combination Therapy Compared With Amlodipine Monotherapy in Hypertensive Patients Uncontrolled on Amlodipine 5 mg Monotherapy
Brief Title: Irbesartan/Amlodipine in Hypertensive Patients Uncontrolled on Amlodipine 5 mg Monotherapy
Acronym: I-COMBINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRBAM_R_04220
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2010-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Irbesartan; Amlodipine

ARMS (2):
- irbesartan/amlodipine (Experimental): Before randomisation : amlodipine 5 mg for 7 to 10 days (common to 2 arms) then After randomisation : irbesartan/amlodipine 150/5 mg fixed combination for 5 weeks followed by irbesartan/amlodipine 150/10 mg fixed combination for 5 additional weeks
  Interventions: Drug: irbesartan/amlodipine
- amlodipine (Active Comparator): Before randomisation : amlodipine 5 mg for 7 to 10 days (common to 2 arms) then After randomisation : amlodipine 5 mg for 5 weeks followed by amlodipine 10 mg for 5 additional weeks
  Interventions: Drug: amlodipine

INTERVENTIONS:
Drug: irbesartan/amlodipine — Pharmaceutical form: 150/5 mg and 150/10 mg tablets (fixed combination) Route of administration: oral Dose regimen: 1 tablet once daily in the morning
  Arms: irbesartan/amlodipine
Drug: amlodipine — Pharmaceutical form: 5 and 10 mg tablets Route of administration: oral Dose regimen: 1 tablet once daily in the morning
  Arms: amlodipine

SUMMARY:
Primary Objective:

* To demonstrate that the antihypertensive efficacy of the fixed combination irbesartan/amlodipine 150/5 mg is superior to that of amlodipine 5 mg monotherapy in lowering systolic blood pressure (SBP) as measured by home blood pressure measurement (HBPM) after 5 weeks of treatment (W5)

Secondary Objective:

* To compare the antihypertensive efficacy of the fixed combination irbesartan/amlodipine 150/5 mg with that of amlodipine 5 mg monotherapy after 5 weeks of treatment (W5)
* To compare the antihypertensive efficacy of the fixed combination therapy irbesartan/amlodipine 150/10 mg with that of amlodipine 10 mg monotherapy at the end of treatment (W10)
* To examine in each treatment group the change from week 5 to week 10 in SBP and diastolic blood pressure (DBP) assessed by HBPM and by office blood pressure measurement (OBPM)
* To determine the incidence and severity of adverse events

ELIGIBILITY:
Inclusion criteria:

* Established essential hypertension
* Treated with amlodipine 5 mg monotherapy for at least 4 weeks
* With uncontrolled BP defined as mean SBP = or > 145 mmHg assessed by OBPM
* Signed written inform consent obtained prior to inclusion in the study

Randomisation Criteria:

* Mean SBP = or > 135 mmHg assessed by HBPM
* Good compliance with the HBPM protocol defined as at least 12 correct measurements performed over the last 6 days of the first period of measurements
* Creatinine clearance = or > 30 ml/min, determined by Cockroft formula

Exclusion criteria:

* Mean SBP = or > 180 mm Hg and/or mean DBP = or > 110 mm Hg measured at doctor's office at Visit 1
* Known or suspected causes of secondary hypertension
* Patients with bilateral artery stenosis, renal artery stenosis in a solitary kidney, renal transplant or only one functioning kidney
* Know contraindications or hypersensitivity to either amlodipine or irbesartan or to the combination or history of angioedema related to the administration of an angiotensin II receptor antagonist or any combination of the drugs used
* Known type 1 diabetes
* Know severe hepatic impairment alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 times the upper limit of normal or history or hepatic encephalopathy, esophageal varices, or portocaval shunt
* Known severe renal impairment (creatinine clearance < 30 ml/mn)
* Concomitant use of any other antihypertensive treatment
* Administration of any other investigational drug within 30 days before inclusion
* Inability to obtain a valid automatic BP measurement recording
* Presence of any severe medical or psychological condition that, in the opinion of the investigator, indicate that participation in the study is not in the best interest of the patient
* Presence of any other conditions (e.g.: geographical, social, etc) that would restrict or limit the patient participation for the duration of the study
* Pregnant or breast feeding women
* Women of childbearing potential unable or unwilling to use an acceptable method to avoid pregnancy for the entire study period

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Mean home systolic blood pressure | At randomisation and week 5

SECONDARY OUTCOMES:
Mean office blood pressure | At randomisation, week 5 and week 10
Mean home diastolic blood pressure | At randomisation, week 5 and week 10

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Genes, MD, Study Director — Sanofi
Locations (40):
- Brazil (8):
  - Sanofi-Aventis Investigational Site Number 07602, Campinas
  - Sanofi-Aventis Investigational Site Number 076-005, Rio de Janeiro
  - Sanofi-Aventis Investigational Site Number 07605, Rio de Janeiro
  - Sanofi-Aventis Investigational Site Number 07604, São José
  - Sanofi-Aventis Investigational Site Number 07601, São Paulo
  - Sanofi-Aventis Investigational Site Number 076-004, São Paulo
  - Sanofi-Aventis Investigational Site Number 076-002, São Paulo
  - Sanofi-Aventis Investigational Site Number 07603, São Paulo
- Chile (5):
  - Sanofi-Aventis Investigational Site Number 15202, Santiago
  - Sanofi-Aventis Investigational Site Number 15203, Santiago
  - Sanofi-Aventis Investigational Site Number 15204, Santiago
  - Sanofi-Aventis Investigational Site Number 15205, Santiago
  - Sanofi-Aventis Investigational Site Number 15206, Santiago
- Colombia (3):
  - Sanofi-Aventis Investigational Site Number 17003, Barranquilla
  - Sanofi-Aventis Investigational Site Number 17004, Barranquilla
  - Sanofi-Aventis Investigational Site Number 17002, Medellín
- Egypt (4):
  - Sanofi-Aventis Investigational Site Number 81803, Alexandria
  - Sanofi-Aventis Investigational Site Number 81804, Alexandria
  - Sanofi-Aventis Investigational Site Number 81801, Cairo
  - Sanofi-Aventis Investigational Site Number 81802, Cairo
- Lebanon (5):
  - Sanofi-Aventis Investigational Site Number 42202, Beirut
  - Sanofi-Aventis Investigational Site Number 42203, Beirut
  - Sanofi-Aventis Investigational Site Number 42204, Beirut
  - Sanofi-Aventis Investigational Site Number 42205, Beirut
  - Sanofi-Aventis Investigational Site Number 42206, Beirut
- Mexico (7):
  - Sanofi-Aventis Investigational Site Number 48401, Durango
  - Sanofi-Aventis Investigational Site Number 48402, Guadalajara
  - Sanofi-Aventis Investigational Site Number 48403, Guadalajara
  - Sanofi-Aventis Investigational Site Number 48406, Guadalajara
  - Sanofi-Aventis Investigational Site Number 48404, Guadalajara
  - Sanofi-Aventis Investigational Site Number 48405, México
  - Sanofi-Aventis Investigational Site Number 48407, México
- Morocco (3):
  - Sanofi-Aventis Investigational Site Number 50401, Casablanca
  - Sanofi-Aventis Investigational Site Number 50402, Marrakesh
  - Sanofi-Aventis Investigational Site Number 50403, Marrakesh
- Tunisia (4):
  - Sanofi-Aventis Investigational Site Number 78804, Aryanah
  - Sanofi-Aventis Investigational Site Number 78803, Monastir
  - Sanofi-Aventis Investigational Site Number 78802, Sfax
  - Sanofi-Aventis Investigational Site Number 78801, Tunis
- Sanofi-Aventis Investigational Site Number 86201, Caracas, Venezuela

REFERENCES:
- [Derived] Bobrie G; I-COMBINE Study Investigators. I-COMBINE study: assessment of efficacy and safety profile of irbesartan/amlodipine fixed-dose combination therapy compared with amlodipine monotherapy in hypertensive patients uncontrolled with amlodipine 5 mg monotherapy: a multicenter, phase III, prospective, randomized, open-label with blinded-end point evaluation study. Clin Ther. 2012 Aug;34(8):1705-19. doi: 10.1016/j.clinthera.2012.06.026. Epub 2012 Jul 30. PMID 22853848